CLINICAL TRIAL: NCT03419260
Title: Electrographic Seizure Management and Neurobehavioral Outcomes in Critically Ill Children
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17-013808; K02NS096058 (NIH)
Record Dates: First submitted 2018-01-24; First posted 2018-02-01 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Seizures
Keywords: seizures; status epilepticus; EEG monitoring
MeSH Terms: conditions — Seizures; Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Critically ill child undergoing clinically indicated EEG monitoring and electrographic seizure management.
  Interventions: Other: Clinically indicated EEG monitoring.

INTERVENTIONS:
Other: Clinically indicated EEG monitoring. — Children enrolled in the study will be undergoing clinically indicated EEG monitoring. Some children will undergo clinically indicated electrographic seizure management.

SUMMARY:
Electrographic seizures are common in critically ill patients leading to increased use of resource-intense continuous EEG monitoring for seizure identification and management. When identified, electrographic seizures are generally treated with anti-seizure medications, but there are very limited data available regarding optimal treatment in terms of the efficacy or safety of specific anti-seizure medications or overall management strategies.

This is a single-center prospective observational study. The investigators aim to: (1) track critically ill patients undergoing clinically indicated EEG monitoring and seizure management to identify risk factors for electrographic seizures, (2) create prediction models guiding EEG monitoring resources to the patients at highest risk for seizures, and (3) evaluate our current management strategy in terms of safety.

DETAILED DESCRIPTION:
Context: Electrographic seizures are common in critically ill patients leading to increased use of resource-intense continuous EEG monitoring for seizure identification and management. When identified, electrographic seizures are generally treated with anti-seizure medications, but there are very limited data available regarding optimal treatment in terms of specific medication selections or overall management strategies. The Children's Hospital of Philadelphia (CHOP) has a formal ICU EEG Monitoring Pathway aiming to standardize EEG monitoring and seizure management. This is a single-center prospective observational study of patients undergoing clinically indicated EEG monitoring to identify risk factors for electrographic seizures and create prediction models guiding limited EEG monitoring resources to the patients at highest risk for seizures, and also to evaluate the current seizure management strategy in terms of safety.

Objectives: The primary objective is to identify risk factors for electrographic seizures in critically ill patients and use these risk factors to create and validate a seizure prediction model. The secondary objective is to evaluate the safety of a targeted and timely electrographic seizure identification and management strategy among critically ill patients guided by a CHOP ICU EEG Monitoring Pathway.

Study Design: Single center observational study of consecutive patients undergoing clinically indicated EEG monitoring.

Setting/Participants: Single-center study of critically ill children in the Pediatric ICU at CHOP undergoing clinically indicated EEG monitoring and seizure management.

ELIGIBILITY:
Inclusion Criteria:

1. Care in the Children's Hospital of Philadelphia Pediatric ICU.
2. Clinically indicated continuous EEG monitoring.
3. Age > 1 month to 18 years.

Exclusion Criteria:

1. Admitted for Phase 2 (intracranial) EEG monitoring.
2. Intensivist expects to discontinue technological support in the next two days given underlying medical or neurological problems.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study is a prospective observational study of consecutive patients undergoing clinically indicated EEG monitoring in the Children's Hospital of Philadelphia Pediatric ICU as guided by an institutional ICU EEG Monitoring Pathway. Each subject will participate from the time of EEG monitoring initiation until the time of hospital discharge. This duration will generally be from several days to several weeks depending on the duration of the hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Electrographic Seizure Occurrence | 3 days
  Percentage of subjects who experience electrographic seizures.

SECONDARY OUTCOMES:
Safety - Mortality | 5 days
  Percentage of subjects with mortality related to electrographic seizure management.
Safety - Occurrence of Cardiopulmonary adverse effects | 5 days
  Percentage of subjects with cardiopulmonary adverse effects related to electrographic seizure management. Cardiopulmonary problems include subcategories of anaphylactic reactions, bradycardia (<5th percentile for age), hypotension (<5th percentile for age), hypoxemia (saturation <90%), lactic acidosis (>2 mmol/l), and intubation requirement.
Safety - Occurrence of Organ Dysfunction | 5 days
  Percentage of subjects with organ dysfunction adverse effects related to electrographic seizure management. Organ dysfunction that will include subcategories of allergic skin manifestations, acute kidney injury, hepatitis and acute liver injury, coagulopathy, and cytopenias (rbc, wbc, platelets).
Safety -Occurrence of Hospital Acquired Infections | 5 days
  Percentage of subjects with hospital acquired infection adverse effects related to electrographic seizure management. Hospital acquired infections that will include subcategories of central line associated bloodstream infections, urinary tract infection, and ventilator associated pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Abend, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fung FW, Jacobwitz M, Vala L, Parikh D, Donnelly M, Xiao R, Topjian AA, Abend NS. Electroencephalographic seizures in critically ill children: Management and adverse events. Epilepsia. 2019 Oct;60(10):2095-2104. doi: 10.1111/epi.16341. Epub 2019 Sep 20. PMID 31538340
- [Background] Fung FW, Jacobwitz M, Parikh DS, Vala L, Donnelly M, Fan J, Xiao R, Topjian AA, Abend NS. Development of a model to predict electroencephalographic seizures in critically ill children. Epilepsia. 2020 Mar;61(3):498-508. doi: 10.1111/epi.16448. Epub 2020 Feb 20. PMID 32077099
- [Background] Fung FW, Parikh DS, Donnelly M, Xiao R, Topjian AA, Abend NS. Electrographic Seizure Characteristics and Electrographic Status Epilepticus Prediction. J Clin Neurophysiol. 2025 Jan 1;42(1):64-72. doi: 10.1097/WNP.0000000000001068. Epub 2024 Jan 9. PMID 38194638
- [Background] Fung FW, Parikh DS, Massey SL, Fitzgerald MP, Vala L, Donnelly M, Jacobwitz M, Kessler SK, Xiao R, Topjian AA, Abend NS. Periodic Discharges in Critically Ill Children: Predictors and Outcome. J Clin Neurophysiol. 2024 May 1;41(4):297-304. doi: 10.1097/WNP.0000000000000986. Epub 2023 Dec 1. PMID 38079254
- [Background] Fung FW, Parikh DS, Donnelly M, Jacobwitz M, Topjian AA, Xiao R, Abend NS. EEG Monitoring in Critically Ill Children: Establishing High-Yield Subgroups. J Clin Neurophysiol. 2024 May 1;41(4):305-311. doi: 10.1097/WNP.0000000000000995. Epub 2023 Mar 8. PMID 36893385
- [Background] Fung FW, Fan J, Parikh DS, Vala L, Donnelly M, Jacobwitz M, Topjian AA, Xiao R, Abend NS. Validation of a Model for Targeted EEG Monitoring Duration in Critically Ill Children. J Clin Neurophysiol. 2023 Nov 1;40(7):589-599. doi: 10.1097/WNP.0000000000000940. Epub 2022 Apr 20. PMID 35512186
- [Background] Fung FW, Parikh DS, Massey SL, Fitzgerald MP, Vala L, Donnelly M, Jacobwitz M, Kessler SK, Topjian AA, Abend NS. Periodic and rhythmic patterns in critically ill children: Incidence, interrater agreement, and seizures. Epilepsia. 2021 Dec;62(12):2955-2967. doi: 10.1111/epi.17068. Epub 2021 Oct 12. PMID 34642942
- [Background] Fung FW, Wang Z, Parikh DS, Jacobwitz M, Vala L, Donnelly M, Topjian AA, Xiao R, Abend NS. Electrographic Seizures and Outcome in Critically Ill Children. Neurology. 2021 May 31;96(22):e2749-e2760. doi: 10.1212/WNL.0000000000012032. PMID 33893203
- [Background] Fung FW, Parikh DS, Jacobwitz M, Vala L, Donnelly M, Wang Z, Xiao R, Topjian AA, Abend NS. Validation of a model to predict electroencephalographic seizures in critically ill children. Epilepsia. 2020 Dec;61(12):2754-2762. doi: 10.1111/epi.16724. Epub 2020 Oct 16. PMID 33063870
- [Background] Fung FW, Fan J, Vala L, Jacobwitz M, Parikh DS, Donnelly M, Topjian AA, Xiao R, Abend NS. EEG monitoring duration to identify electroencephalographic seizures in critically ill children. Neurology. 2020 Sep 15;95(11):e1599-e1608. doi: 10.1212/WNL.0000000000010421. Epub 2020 Jul 20. PMID 32690798